CLINICAL TRIAL: NCT03998423
Title: Oral Fecal Microbiota Transplant Feasibility Study in Alzheimer's Disease
Acronym: AMBITION
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: SARS-CoV-2 has been detected in fecal material. Although FMT is screened for SARS-CoV-2, the team decided to end the study to minimize risk to participants.
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wisconsin Partnership Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMBITION; 2018-0283 (Other: UW IRB); A534255 (Other: UW Madison); SMPH/MEDICINE/MEDICINE (Other: UW Madison)
Record Dates: First submitted 2018-08-23; First posted 2019-06-26 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: A single dose of 30 capsules (22.5g) of oral FMT will be given once (week 0), twice (week 0 and week 8), or three times (week 0, week 8, and week 24). Participants are randomly assigned to 1, 2, or 3 doses of FMT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 dose fecal microbiota transplant (Experimental): This group will receive one dose of Fecal Microbiota Transplant (FMT) at baseline.
  Interventions: Biological: Fecal Microbiota Transplant
- 2 doses fecal microbiota transplant (Experimental): This group will will receive one dose of Fecal Microbiota Transplant (FMT) at baseline and a second dose of FMT 8 weeks later.
  Interventions: Biological: Fecal Microbiota Transplant
- 3 doses fecal microbiota transplant (Experimental): This group will will receive one dose of Fecal Microbiota Transplant (FMT) at baseline, second dose of FMT at 8 weeks, and a third dose of FMT at 12 weeks.
  Interventions: Biological: Fecal Microbiota Transplant

INTERVENTIONS:
Biological: Fecal Microbiota Transplant — Double-encapsulated Fecal Microbiota Transplant Capsules
  Other Names: FMT Capsule DE

SUMMARY:
The goal of this study is to assess the safety and feasibility of an oral fecal microbiota transplant (FMT) intervention for Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Studies suggests that microbes, including those derived from the gut, may play a role in the development or progression of AD. Gut microbiome composition among individuals with the Alzheimer's clinical syndrome is reduced in microbial diversity and shows compositional differences relative to control groups. Further, genera identified as more abundant in AD are associated with greater AD pathology while genera identified as less abundant in AD are associated with less AD pathology, as shown using CSF biomarkers.

The goal of this study is to assess the safety and feasibility of an oral fecal microbiota transplant (FMT) intervention.

* Primary Objective: To assess the safety and feasibility (recruitment, eligibility, enrollment, completion, and follow-up) of an oral FMT intervention in people with and without the Alzheimer's clinical syndrome.
* Secondary Objective: To demonstrate the effects of FMT on the composition and function of the gut microbiota. To collect preliminary data in order to estimate sample size and other parameters for a larger study.

ELIGIBILITY:
Inclusion Criteria:

* Current enrollment in the Wisconsin ADRC clinical core study (2011-0030), ADCP (26695, MCW IRB), or referred from clinic
* At least 45 years of age
* Good general health (other than dementia) with no conditions/medications affecting the gut microbiome (see exclusion criteria below)
* Willing and able to comply with all study procedures for the duration of the study
* Able to provide signed and date informed consent form
* Participant is not pregnant, lactating or of childbearing potential (ie women must be two years post-menopausal or surgically sterile
* Males must agree to avoid impregnation of women during and for four weeks after completing study treatment through use of an acceptable method of contraception
* Able to take oral medications
* Able to take the test capsule successfully with no signs or symptoms of dysphagia

Additional inclusion criteria for participants with Alzheimer's disease:

* Abnormal memory function documented by neuropsychological testing
* Wisconsin ADRC (HS IRB# 2015-0030) Consensus Diagnosis Conference indicates probable AD diagnosis as per NINDS/ADRDA criteria for probable AD (for ADRC and ADCP participants only).

Exclusion Criteria:

* Active or previous (within 6 months) participation in an Alzheimer's clinical intervention/trial
* Significant neurologic disease: Any significant neurologic disease, such as Parkinson's disease, stroke, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, subdural hematoma, multiple sclerosis, seizure disorder, or other significant deficits (other than Alzheimer's dementia)
* Alcohol/substance: history of alcohol/substance dependence since joining the cohort
* Psychiatric disorders: Untreated current axis 1 DSM-V disorder such as major untreated depression, current untreated bipolar 1 disorder, untreated schizophrenia spectrum disorders, or other conditions potentially affecting study adherence.
* Significant medical illness: any significant systemic illness or unstable medical condition occurring that could affect cognition (other than Alzheimer's). Examples include malignant cancer, chemotherapy, untreated thyroid disease, heart failure, or renal insufficiency.
* Illiterate, blind, or non-English speaking
* Known periodic antibiotic use (i.e. prior to dental appointments)
* Oral FMT-specific exclusion criteria:

  * Inability (e.g. dysphagia) or unwilling to swallow capsules - assessed using the Eating Assessment Tool (EAT-10) and bedside 3oz water swallow test administered by CRU nurse or study coordinator
  * Active gastrointestinal infection at time of enrollment
  * Known or suspected toxic megacolon and/or known small bowel ileus
  * History of total colectomy or bariatric surgery
  * Concurrent intensive induction chemotherapy, radiation therapy, or biological treatment for active malignancy
  * Unable or unwilling to comply with protocol requirements
  * Expected life expectancy < 6 months
  * Previous FMT or microbiome-based products at any time excluding this study
  * Patients with severe anaphylactic or anaphylactoid food allergy
  * Solid organ transplant recipients ≤ 90 days post-transplant or on active treatment for rejection
  * Immunocompromised/ at risk of CMV/EBV associated disease
  * A condition that would jeopardize the safety or rights of the subject, would make it unlikely for the subject to complete the study, or would confound the results of the study
* Exclusionary factors affecting the microbiome:

  * Use of systemic antibiotics (intravenous, intramuscular, or oral) in the previous 3 months
  * Oral, intravenous, intramuscular, nasal or inhaled corticosteroids (except PRN use for allergies)
  * Immune stimulating medications
  * Methotrexate or immunosuppressive cytotoxic agents
  * Large doses of commercial probiotics consumed (greater than or equal to 108 cfu or organisms per day). Includes tablets, capsules, lozenges, chewing gum or powders in which probiotic is a primary component (ordinary dietary components such as fermented beverages/milks, yogurts, foods do not apply).
  * Unstable dietary history during the previous month, which is defined as major changes in diet by eliminating or significantly increasing a major good group
  * Major surgery of the GI tract, with the exception of cholecystectomy and appendectomy, in the past five years
  * Major bowel resection at any time
  * Active uncontrolled gastrointestinal disorders or disease including: inflammatory bowel disease including ulcerative colitis (mild-moderate-severe), Crohn's disease (mild-moderate-severe), or indeterminate colitis; irritable bowel syndrome (moderate-severe); persistent, infectious gastroenteritis, colitis or gastritis; persistent or chronic diarrhea of unknown etiology, Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated), or chronic constipation

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Safety: Proportion of participants with treatment-related adverse events, serious adverse events, or adverse events of special interest. | 1 year
  Proportion of participants with treatment-related adverse events, serious adverse events, or adverse events of special interest.
  Adverse events, serious adverse events, or adverse events of special interest, will be evaluated following study procedures using AE and SAE forms, telephone and in person interview, and relevant medical records related to adverse events.
Feasibility: Participant recruitment rate | 1 year
  Number of weeks/months needed to meet study group numbers.
Feasibility: Eligibility | 1 year
  Proportion of individuals expressing interest who meet inclusion/exclusion criteria.
Feasibility: Procedures completed. | 1 year
  Proportion of participants able to complete procedures (including FMT) will be part of feasibility.
Feasibility: Retention | 1 year
  Proportion of participants that complete follow up.
Change in gut composition: Engraftment of fecal microbial transplant as assessed by 16S rRNA sequencing of recipient stool sample | baseline, 8 weeks, 24 weeks, 1 year
  In order to determine efficacy of fecal transplant, change in composition, i.e. microbial engraftment will be assessed by testing for newly detected operational taxonomic units (OTUs) in the gut microbiome of a participant post-FMT (which were present in the donor but undetected in the participant pre-FMT). This will be assessed via 16S rRNA seq of recipient stool samples pre- and post- FMT.

SECONDARY OUTCOMES:
Cognition: Change in Montreal Cognitive Assessment (MoCA) score | baseline and 1 year
  The Montreal Cognitive Assessment (MoCA) is a cognitive screening test used for detecting cognitive impairment. MoCA scores range between 0 and 30. Lower scores are indicative of impairment
Cognition: Change in results of Repeatable Battery for the Assessment of Neuropsychological Status | baseline and 1 year
  The Repeatable Battery for the Assessment of Neuropsychological Status consists of twelve subtests which give five scores, one for each of the five domains tested (immediate memory, visuospatial/constructional, language, attention, delayed memory). Raw scores on each domain are scaled to account for a person's age. Scaled scores are converted to percentiles which are used to determine a range of performance (impaired, borderline impaired, expected score, high average, superior) and overall cognitive status (impaired/not impaired).
Cognition: Change in the results of Trail Making Test Part A and Part B | baseline and 1 year
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts, A and B. Participant is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning.
  Results for both TMT A and B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
Metabolic/physiological measure: Change in the level of Hemoglobin A1C | baseline, 8 weeks, 24 weeks, and 1 year
  Change in the level of Hemoglobin A1C will be assessed
Metabolic/physiological measure: Change in the level of fasting glucose | baseline, 8 weeks, 24 weeks, and 1 year
  Change in the level of fasting glucose will be assessed
Metabolic/physiological measure: Change in the level of fasting insulin | baseline, 8 weeks, 24 weeks, and 1 year
  Change in the level of fasting insulin will be assessed
Metabolic/physiological measure: Change in the level of C-reactive protein | baseline, 8 weeks, 24 weeks, and 1 year
  Change in the level of C-reactive protein will be assessed
Metabolic/physiological measure: Change in the blood lipid profile | baseline, 8 weeks, 24 weeks, and 1 year
  Change in the blood lipid profile will be assessed
Metabolic/physiological measure: Change in the blood pressure | baseline, 8 weeks, 24 weeks, and 1 year
  Change in the blood pressure will be assessed
Metabolic/physiological measure: Change in body weight | baseline, 8 weeks, 24 weeks, and 1 year
  Change in body weight will be assessed
Metabolic/physiological measure: Change in the body composition by measuring body fat percentage | baseline and 1 year
  Change in the body composition by measuring body fat percentage
Change in insulin resistance indexed by the homeostatic model assessment-insulin resistance (HOMA-IR) method | baseline, 8 weeks, 24 weeks, and 1 year
  Fasting glucose and fasting insulin will be used to calculate HOMA-IR.
Change in physical activity as measured by Actigraphy watch | baseline, 24 weeks, and 1 year
  Actigraphy watch will be worn on the non-dominant wrist was used to record a participant's physical activity (total number of active minutes per day).
Change in Sleep as measured by Actigraphy watch | baseline, 24 weeks, and 1 year
  Actigraphy watch will be worn on the non-dominant wrist to estimate sleep duration.
Change in CSF biomarkers | baseline and 1 year
  Aβ42, Aβ42/Aβ40, phosphorylated tau, total tau, YKL-40
Change in serum/plasma metabolites on an average of one week pre and post FMT | baseline, week 8, week 24, and 1 year
  Change in serum/plasma metabolites on an average of one week pre and post FMT
Function: Change in total score on the Bristol Activities of Daily Living Scale | baseline and 1 year
  Change in total score on the Bristol Activities of Daily Living Scale. This is a tool used to measure functional ability (ability to independently carry out activities of daily living), and was developed for use with people with dementia. The minimum score is "0". The maximum score is "60". A lower score (better) indicates that a person is independent in their activities of daily living, and a higher score (worse) indicates that the individual is dependent on others.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Bendlin, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vogt NM, Kerby RL, Dill-McFarland KA, Harding SJ, Merluzzi AP, Johnson SC, Carlsson CM, Asthana S, Zetterberg H, Blennow K, Bendlin BB, Rey FE. Gut microbiome alterations in Alzheimer's disease. Sci Rep. 2017 Oct 19;7(1):13537. doi: 10.1038/s41598-017-13601-y. PMID 29051531